CLINICAL TRIAL: NCT04858035
Title: Online Assessment and Enhancement of Auditory Perception for Speech Sound Errors: Online Perceptual Training for RSE
Brief Title: Auditory-Perceptual Training Via Telepractice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montclair State University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); Syracuse University (Other); New York University (Other)
Responsible Party: Principal Investigator, Elaine Hitchcock, Associate Professor, Montclair State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-21-2137-Study 3; R15DC019775-01 (NIH)
Record Dates: First submitted 2021-04-05; First posted 2021-04-26 (Actual); Results first posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Speech Sound Disorder
Keywords: speech sound disorder; auditory perception; articulation
MeSH Terms: conditions — Speech Sound Disorder

STUDY DESIGN:
Intervention Model Description: This study follows a multiple-baseline across-subjects design with random assignment of participants to different baseline durations. Following the initial evaluation to determine eligibility, participants will be enrolled in a baseline phase in which perception and production abilities will be probed but not treated. Perception will be measured using the online identification and category goodness tasks and production will be measured from standard probes containing /r/ in various phonetic contexts. Participants will be randomly assigned to transition from the baseline to the treatment condition at one of 7 possible points, ranging from 3 to 9 baseline sessions. All participants will receive 12 sessions of perceptual training over 4 weeks followed by 4 sessions of production training over 2 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Online Speech Training (Experimental): Participants will be randomly assigned to transition from the baseline to the treatment condition at one of 7 possible points, ranging from 3 to 9 baseline sessions. All participants will receive 12 sessions of perceptual training over 4 weeks. Finally, participants will complete a 3-session maintenance phase in which perception and production are probed but not treated. Perception will be measured using the identification and category goodness judgment.
  Following completion of perception training all participants will complete two weeks of production training. The production training will consists of 4, 60-minute sessions. Each session will provide instruction and practice trials.
  Interventions: Behavioral: Perceptual training; Behavioral: Production training

INTERVENTIONS:
Behavioral: Perceptual training — Perceptual training involves self-paced presentation of auditory stimuli via a computerized software program.
  Stimuli are organized into three separate tasks:
  Tasks 1 and 3 will train category goodness judgment: Participants will hear 75 naturally produced speech tokens containing /r/ from various speakers, with a balance of correct and incorrect productions. They will classify each /r/ as correct or incorrect and receive feedback on the accuracy of their classification. Tasks 1 and 3 differ in that task 1 will feature a subset of items designed to provide focused practice on a specific context (e.g., initial /r/ as in red; /r/ as syllable nucleus as in sir), with increasing difficulty over time, whereas task 3 will feature randomly selected items representing all contexts and difficulty levels.
  Task 2: Participants will hear 75 items drawn from the synthetic rake-wake continuum used in the identification task administered at baseline.
Behavioral: Production training — Instruction: Discuss tongue shapes for /r/. Pre-practice: relatively unstructured, highly interactive elicitation; provide models and placement cue and KP on every trial.
  Structured syllable practice: Practice will occur in blocks of 10 consecutive trials on the same syllable (e.g., 10 /ra/), after which a new syllable will be addressed (e.g., 10 /re/--but note that in the fully blocked condition, the same syllable should occur in two consecutive blocks of 10).

SUMMARY:
The objective of this study is to measure the effects of online perceptual training on perception and production in children with RSE who exhibit atypical perception relative to norms from our lab-based pilot data. In a multiple-baseline across-subjects design, 10 children with RSE will begin in a baseline phase probing perceptual acuity for /r/. Perceptual training with multiple types of stimuli will be initiated in a staggered fashion. Production probes elicited before and after treatment will assess the extent to which perception gains transfer to /r/ production.

DETAILED DESCRIPTION:
Following the initial evaluation to determine eligibility, participants will be enrolled in a baseline phase in which perception and production abilities will be probed but not treated. In a multiple-baseline across-subjects design with randomization, the 10 participants will be randomly assigned to transition from the baseline to the treatment condition at one of 7 possible points, ranging from 3 to 9 baseline sessions. After baseline sessions, perceptual training will be delivered in twelve 30-minute sessions occurring 3 times per week for 4 weeks. The training is fully computerized and can be self-administered, but a study clinician will attend one session per participant per week to ensure attention to study tasks. Each session will feature three listening tasks of approximately equal duration. Following perceptual training, participants will receive 4 60-minute sessions of production training completed over two weeks.

ELIGIBILITY:
Inclusion Criteria:

* Must be between 9;0 and 15;11 years of age at the time of enrollment.
* Must speak English as the dominant language (i.e., must have begun learning English by age 2, per parent report).
* Must speak a rhotic dialect of English.
* Must pass a pure-tone hearing screening at 20dB HL
* Must pass a brief examination of oral structure and function.
* Must exhibit less than 30% accuracy, based on consensus across 2 trained listeners, on a probe list eliciting rhotics in various phonetic contexts at the word level.
* Must exhibit no more than 3 sounds other than /r/ in error on the GFTA-3

Exclusion Criteria:

* Must not receive a T score more than 1.3 SD below the mean on the Wechsler Abbreviated Scale of Intelligence-2 (WASI-2) Matrix Reasoning
* Must not receive a scaled score of 7 or higher on the Recalling Sentences and Formulated Sentences subtests of the Clinical Evaluation of Language Fundamentals-5 (CELF-5).
* Must not have an existing diagnosis of developmental disability or major neurobehavioral syndrome such as cerebral palsy, Down Syndrome, or Autism Spectrum Disorder

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elaine R. Hitchcock, PhD, Principal Investigator — Montclair State University
Locations (1):
- Montclair State University- Online Research Study, Upper Montclair, New Jersey, United States

REFERENCES:
- [Background] Preston JL, Hitchcock ER, Leece MC. Auditory Perception and Ultrasound Biofeedback Treatment Outcomes for Children With Residual /ɹ/ Distortions: A Randomized Controlled Trial. J Speech Lang Hear Res. 2020 Feb 26;63(2):444-455. doi: 10.1044/2019_JSLHR-19-00060. Epub 2020 Feb 26. PMID 32097058
- [Background] Byun TM, Hitchcock ER. Investigating the use of traditional and spectral biofeedback approaches to intervention for /r/ misarticulation. Am J Speech Lang Pathol. 2012 Aug;21(3):207-21. doi: 10.1044/1058-0360(2012/11-0083). Epub 2012 Mar 21. PMID 22442281
- [Background] McAllister Byun T. Efficacy of Visual-Acoustic Biofeedback Intervention for Residual Rhotic Errors: A Single-Subject Randomization Study. J Speech Lang Hear Res. 2017 May 24;60(5):1175-1193. doi: 10.1044/2016_JSLHR-S-16-0038. PMID 28389677
- [Background] McAllister Byun T, Harel D, Halpin PF, Szeredi D. Deriving gradient measures of child speech from crowdsourced ratings. J Commun Disord. 2016 Nov-Dec;64:91-102. doi: 10.1016/j.jcomdis.2016.07.001. Epub 2016 Jul 6. PMID 27481555
- [Background] Harel D, Hitchcock ER, Szeredi D, Ortiz J, McAllister Byun T. Finding the experts in the crowd: Validity and reliability of crowdsourced measures of children's gradient speech contrasts. Clin Linguist Phon. 2017;31(1):104-117. doi: 10.3109/02699206.2016.1174306. Epub 2016 Jun 7. PMID 27267258
- [Background] Preston JL, Benway NR, Leece MC, Hitchcock ER, McAllister T. Tutorial: Motor-Based Treatment Strategies for /r/ Distortions. Lang Speech Hear Serv Sch. 2020 Oct 2;51(4):966-980. doi: 10.1044/2020_LSHSS-20-00012. Epub 2020 Aug 12. PMID 32783706
- [Background] Byun TM, Hitchcock ER, Swartz MT. Retroflex versus bunched in treatment for rhotic misarticulation: evidence from ultrasound biofeedback intervention. J Speech Lang Hear Res. 2014 Dec;57(6):2116-30. doi: 10.1044/2014_JSLHR-S-14-0034. PMID 25088034
- [Background] Dugan SH, Silbert N, McAllister T, Preston JL, Sotto C, Boyce SE. Modelling category goodness judgments in children with residual sound errors. Clin Linguist Phon. 2019;33(4):295-315. doi: 10.1080/02699206.2018.1477834. Epub 2018 May 24. PMID 29792525
- [Background] McAllister Byun T, Tiede M. Perception-production relations in later development of American English rhotics. PLoS One. 2017 Feb 16;12(2):e0172022. doi: 10.1371/journal.pone.0172022. eCollection 2017. PMID 28207800
- [Background] McAllister T, Preston JL, Hitchcock ER, Hill J. Protocol for Correcting Residual Errors with Spectral, ULtrasound, Traditional Speech therapy Randomized Controlled Trial (C-RESULTS RCT). BMC Pediatr. 2020 Feb 11;20(1):66. doi: 10.1186/s12887-020-1941-5. PMID 32046671
- [Background] Hitchcock ER, Byun TM. Enhancing generalisation in biofeedback intervention using the challenge point framework: a case study. Clin Linguist Phon. 2015 Jan;29(1):59-75. doi: 10.3109/02699206.2014.956232. Epub 2014 Sep 12. PMID 25216375
- [Background] McAllister Byun T, Swartz MT, Halpin PF, Szeredi D, Maas E. Direction of attentional focus in biofeedback treatment for /r/ misarticulation. Int J Lang Commun Disord. 2016 Jul;51(4):384-401. doi: 10.1111/1460-6984.12215. Epub 2016 Mar 6. PMID 26947142
- [Background] Hitchcock, ER, Cabbage, KL, Swartz, M, Carrell, T. Measuring Speech Perception Using the Wide-Range Acoustic Accuracy Scale: Preliminary Findings. Perspectives of the ASHA Special Interest Groups, 5(4):1098-1112, 2020.
- [Background] Hitchcock ER, Swartz MT, Lopez M. Speech Sound Disorder and Visual Biofeedback Intervention: A Preliminary Investigation of Treatment Intensity. Semin Speech Lang. 2019 Mar;40(2):124-137. doi: 10.1055/s-0039-1677763. Epub 2019 Feb 22. PMID 30795023
- [Background] Byun TM, Hitchcock ER, Ferron J. Masked Visual Analysis: Minimizing Type I Error in Visually Guided Single-Case Design for Communication Disorders. J Speech Lang Hear Res. 2017 Jun 10;60(6):1455-1466. doi: 10.1044/2017_JSLHR-S-16-0344. PMID 28595354
- [Background] Hitchcock ER, Harel D, Byun TM. Social, Emotional, and Academic Impact of Residual Speech Errors in School-Aged Children: A Survey Study. Semin Speech Lang. 2015 Nov;36(4):283-94. doi: 10.1055/s-0035-1562911. Epub 2015 Oct 12. PMID 26458203

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were enrolled between January 21, 2022 and July 30, 2024. All participants were assessed and treated online using standardized headphones which were mailed to them prior to the onset of the study.
Pre-assignment Details: No significant events were encountered over the course of this study.
Groups:
- Online Speech Perception Training: Participants will be randomly assigned to transition from the baseline to the treatment condition at one of 7 possible points, ranging from 3 to 9 baseline sessions. All participants will receive 12 sessions of perceptual training over 4 weeks. Finally, participants will complete a 3-session maintenance phase in which perception and production are probed but not treated. Perception will be measured using the identification and category goodness judgment.
  Following completion of perception training all participants will complete two weeks of production training. The production training will consists of 4, 60-minute sessions. Each session will provide instruction and practice trials.
Period: Overall Study
Arm/Group | Online Speech Perception Training
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Online Speech Perception Training: Participants will be randomly assigned to transition from the baseline to the treatment condition. All participants will complete the assigned # of baselines sessions in which perception and production probes are elicited. All participants will then receive 12 sessions of perceptual training over 4 weeks, followed by 4 stimulability production training sessions. Participants will complete a 3-session maintenance phase in which perception and production are probed but not treated.
Arm/Group | Online Speech Perception Training
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 1
  Unknown or Not Reported | 0
Percent Accuracy Perception Task [Mean (Standard Deviation); unit: percent accuracy] — Prior to any perception training, participants will listen recordings of single words containing /r/ in various word positions one at a time and will be cued to rate the /r/ in each production as correct or incorrect. Performance will be quantified as percent agreement with expert listeners and reported here as an average baseline level of function prior to any perceptual training tasks..
  percent accuracy | 1.84 (0.97)
Perceptually Rated Accuracy of /r/ Word Production [Mean (Standard Deviation); unit: percent accuracy] — Prior to any perception or speech production training, participants will complete standard word probes containing /r/ in various phonetic context.
  percent accuracy | 5.87 (1.28)

OUTCOME MEASURES:

1. Primary Outcome: Averaged Perception Percent Accuracy Score
Description: Averaged percent accuracy post-perception training.
Time Frame: Participants' perception progress was tracked across all treatment phases. The averaged percent accuracy score reported here was collected during maintenance sessions (3 sessions across 1 week).
Measure: Mean (Standard Deviation); unit: percent accuracy
Groups:
- Online Speech Perception Training: Participants will be randomly assigned to transition from the baseline to the treatment condition. All participants will receive 12 sessions of perceptual training over 4 weeks, followed by 1 training and 3 stimulability production training sessions. Participants will complete a 3-session maintenance phase in which perception and production are probed but not treated.
Arm/Group | Online Speech Perception Training
Number analyzed (Participants) | 10
percent accuracy | 84.74 (9.53)

2. Secondary Outcome: Raw Change in Percent Accuracy Perception Task
Description: Represents the raw change in percent accuracy on the perception task, calculated as the difference between the average pre-training accuracy score and the average post-training accuracy score.
Time Frame: Participants' progress was tracked across pre-treatment phase (averaged baselines) compared to post treatment phase (averaged three maintenance sessions which occurred over 1 week), up to 8 weeks, including baselines, treatment, and maintenance sessions.
Measure: Mean (Full Range); unit: percent accuracy
Groups:
- Online Speech Perception Training: Participants will be randomly assigned to transition from the baseline to the treatment condition. All participants will receive 12 sessions of perceptual training over 4 weeks, a midpoint assessment, f 4 sessions of production training, and a 3-session maintenance phase.
  Tasks 1 and 3 will train category goodness judgment: Participants will hear 75 naturally produced speech tokens containing /r/ from various speakers, with a balance of correct and incorrect productions. They will classify each /r/ as correct or incorrect and receive feedback on the accuracy of their classification. Tasks 1 and 3 differ in that task 1 will feature a subset of items designed to provide focused practice on a specific context (e.g., initial /r/ as in red; /r/ as syllable nucleus as in sir), with increasing difficulty over time, whereas task 3 will feature randomly selected items representing all contexts and difficulty levels.
  Task 2: Participants will hear 75 items drawn from the synthetic rake-wake continuum used in the identification task administered at baseline.
  Production training: Instruction: Discuss tongue shapes for /r/. Pre-practice: relatively unstructured, highly interactive elicitation; with models and cueing per trial.
  Structured syllable practice: Practice will occur in blocks of 10 consecutive trials on the same syllable (e.g., 10 /ra/), after which a new syllable will be addressed (e.g., 10 /re/.
Arm/Group | Online Speech Perception Training
Number analyzed (Participants) | 10
percent accuracy | 10.57 [5.34 to 20.33]

3. Secondary Outcome: Perceptually Rated Accuracy of /r/ Word Production
Description: Perceptually rated accuracy of /r/ word production probes across an average of four expert listeners post perception and production training.
Time Frame: as for outcome 2
Measure: Mean (Full Range); unit: percent accuracy
Groups:
- Online Perception Speech Training: Participants will be randomly assigned to transition from the baseline to the treatment condition at one of 7 possible points, ranging from 4 to 10 baseline sessions. All participants will receive 12 sessions of perceptual training over 4 weeks. Finally, participants will complete a 3-session maintenance phase in which perception and production are probed but not treated. Perception will be measured using the identification and category goodness judgment.
Arm/Group | Online Perception Speech Training
Number analyzed (Participants) | 10
percent accuracy | 23.45 [-1.88 to 50.55]

ADVERSE EVENTS:
Time Frame: 4 months
Description: Participants were surveyed in post treatment assessment sessions where they asked if they experienced any discomfort or side effects from the treatment.
Groups:
- Online Speech Perception Training: Participants will be randomly assigned to transition from the baseline to the treatment condition at one of 7 possible points, ranging from 4 to 10 baseline sessions. All participants will receive 12 sessions of perceptual training over 4 weeks. Finally, participants will complete a 3-session maintenance phase in which perception and production are probed but not treated. Perception will be measured using the identification and category goodness judgment.
  Following completion of perception training all participants will complete two weeks of production training. The production training will consists of 4, 60-minute sessions. Each session will provide instruction and practice trials.
Arm/Group | Online Speech Perception Training
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2020-10-21): https://cdn.clinicaltrials.gov/large-docs/35/NCT04858035/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-17): https://cdn.clinicaltrials.gov/large-docs/35/NCT04858035/SAP_001.pdf
  • Informed Consent Form (2022-02-09): https://cdn.clinicaltrials.gov/large-docs/35/NCT04858035/ICF_002.pdf